CLINICAL TRIAL: NCT00001366
Title: MRI-Based Functional Language Mapping in Children With Epilepsy
Brief Title: Mapping the Areas of the Brain Associated With Language in Children With Epilepsy
Status: Completed | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 930191; 93-N-0191
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2002-09

CONDITIONS: Epilepsy; Seizures
Keywords: Neuroimaging; Seizures; Cerebral Localization; Partial Epilepsy; Epilepsy
MeSH Terms: conditions — Epilepsy; Seizures; Epilepsies, Partial

SUMMARY:
Researchers are interested in studying if magnetic resonance imaging (MRI) is practical for locating the areas of the brain associated with language in children with epilepsy.

When a region of the brain is active, it uses more fuel in the form of oxygen and sugar (glucose). As the brain uses more fuel it produces more waste products, carbon dioxide and water. Blood carries fuel to the brain and waste products away from the brain. As brain activity increases blood flow to and from the area of activity increases also.

Patients participating in the study will be asked to perform tasks designed to test language skills while undergoing an MRI to detect areas of the brain using oxygen and receiving blood flow.

DETAILED DESCRIPTION:
We propose to study the feasibility of utilizing MRI to perform functional mapping of language cortex in children with epilepsy. We will use 1.5 Tesla MRI to study cerebral blood flow and tissue oxygenation during cognitive activation tasks derived from previous adult studies.

ELIGIBILITY:
Children aged 5-17 years.

Partial epilepsy (localized).

Ability to cooperate with task paradigms (IQ greater than 65).

No cardiac pacemakers, cochlear implants, shrapnel, vascular clips, braces, or claustrophobia.

No one with inability to cooperate with task paradigms.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 230
Dates: Start 1993-08; Study Completion 2002-09

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Neurological Disorders and Stroke (NINDS), Bethesda, Maryland, United States

REFERENCES:
- [Background] Hertz-Pannier L, Gaillard WD, Mott SH, Cuenod CA, Bookheimer SY, Weinstein S, Conry J, Papero PH, Schiff SJ, Le Bihan D, Theodore WH. Noninvasive assessment of language dominance in children and adolescents with functional MRI: a preliminary study. Neurology. 1997 Apr;48(4):1003-12. doi: 10.1212/wnl.48.4.1003. PMID 9109891
- [Background] Bookheimer SY, Zeffiro TA, Blaxton T, Malow BA, Gaillard WD, Sato S, Kufta C, Fedio P, Theodore WH. A direct comparison of PET activation and electrocortical stimulation mapping for language localization. Neurology. 1997 Apr;48(4):1056-65. doi: 10.1212/wnl.48.4.1056. PMID 9109900
- [Background] Malow BA, Blaxton TA, Sato S, Bookheimer SY, Kufta CV, Figlozzi CM, Theodore WH. Cortical stimulation elicits regional distinctions in auditory and visual naming. Epilepsia. 1996 Mar;37(3):245-52. doi: 10.1111/j.1528-1157.1996.tb00020.x. PMID 8598182